CLINICAL TRIAL: NCT06782373
Title: PAXIS: A Randomized, Double-blind, Placebo-controlled Dose-finding Phase 2 Study (Part 1) Followed by an Open-label Period (Part 2) to Assess the Efficacy and Safety of Pacritinib in Patients With VEXAS Syndrome
Brief Title: A Study to Assess the Effectiveness and Safety of Pacritinib in Patients With VEXAS Syndrome (PAXIS)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: PSI CRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PAC601; 2024-516347-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-07; First posted 2025-01-17 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: VEXAS; VEXAS Syndrome
Keywords: Vacuoles; E1 Ubiquitin-activating enzyme; X-linked; Autoinflammatory; Somatic syndrome; UBA1; Hematologic neoplasms; Myelodysplastic Syndromes; Pacritinib; Myeloid progenitors
MeSH Terms: conditions — VEXAS syndrome; Hematologic Neoplasms; Myelodysplastic Syndromes | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1:1 to receive pacritinib dose A, pacritinib dose B plus placebo, or placebo for up to 24 weeks during a double-blind treatment period, followed by treatment with pacritinib during an open-label treatment period for up to 48 weeks. Randomization will be stratified by prescribed GC dose on the day of randomization.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In the double-blind portion of the trial, the Sponsor, trial participants, and Investigators will be blinded to treatment assignments. Active and placebo products will be of identical appearance. The Independent Data Monitoring Committee will have access to unblinded data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pacritinib (Experimental): To receive oral administration of pacritinib dose A for up to 24 weeks.
  Interventions: Drug: Pacritinib
- Pacritinib + placebo (Experimental): To receive oral administration of pacritinib dose B plus placebo for up to 24 weeks
  Interventions: Drug: Pacritinib; Drug: Placebo
- Placebo (Placebo Comparator): To receive oral administration of placebo for up to 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pacritinib — Supplied in hard capsules.
  Arms: Pacritinib; Pacritinib + placebo
Drug: Placebo — Supplied in hard capsules.
  Arms: Pacritinib + placebo; Placebo

SUMMARY:
This trial is to assess the effectiveness and safety of pacritinib in patients with VEXAS (i.e., Vacuoles in myeloid progenitors, E1 ubiquitin-activating enzyme, X-linked, autoinflammatory manifestations, and somatic) syndrome. 78 participants will be enrolled, randomized to either pacritinib dose A, pacritinib dose B + placebo, or placebo. Randomization will be stratified by prescribed GC dose on the day of randomization.

DETAILED DESCRIPTION:
This trial is a randomized, multicenter, double-blind, placebo-controlled phase 2 trial (Part 1) followed by an open-label treatment period (Part 2) designed to evaluate the efficacy and safety of pacritinib for the prevention of VEXAS flares after glucocorticoid (GC) taper. The trial will enroll participants ≥18 years with inflammatory VEXAS syndrome receiving ongoing GC therapy for ≥4 consecutive weeks, requiring between 15 and 45 mg daily (of prednisone / prednisolone or equivalent) at the time of enrollment (randomization). Participants will be randomized 1:1:1 to receive pacritinib dose A (n=26), pacritinib dose B plus placebo (n=26), or placebo (n=26) for up to 24 weeks during a double-blind treatment period, followed by treatment with pacritinib during an open-label treatment period for up to 48 weeks. Participants who complete the open-label treatment period at End of Week (EOW) 48 and who are benefitting from pacritinib in the opinion of the Investigator may continue to receive treatment for an additional 1 year on the extension period. Participants who discontinue study treatment will have a 30-day post-End of Treatment (EOT) follow-up period. Randomization will be stratified by prescribed GC dose on the day of randomization. All outcomes will be reported by treatment arm, and pair-wise comparison between each pacritinib arm and placebo will be performed in the double-blind treatment period.

Participants who complete the double-blind treatment period at EOW 24 or meet Early Failure criteria at EOW 12 will transition to an open-label pacritinib treatment period through EOW 48. In addition, if a trial arm closes due to interim futility or safety, all participants currently randomized to that arm will transition to open-label treatment.

The trial (including the double-blind and open-label treatment periods, as well as the extension period) is planned to end approximately 2 years from the first dose of the last participant.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented evidence of a pathogenic mutation at methionine-41 (M41) or neighboring splice site mutation (c.118-1, c.118-2) position in UBA1 mutation based on myeloid next-generation sequencing (NGS) droplet digital polymerase chain reaction (ddPCR), or Sanger sequencing in peripheral blood or bone marrow samples.
* Current or documented evidence of past inflammatory involvement within 6 months prior to enrollment of at least one of the following organ systems by VEXAS syndrome: cutaneous (e.g., neutrophilic dermatosis, cutaneous vasculitis), vasculature (e.g., vasculitis), musculoskeletal (e.g., chondritis, arthritis), ocular (e.g., uveitis, scleritis), periorbital (e.g. periorbital edema), genitourinary (e.g., epididymitis), or pulmonary (e.g., alveolitis).
* Receiving ongoing GC therapy (stable prednisone or prednisolone dose of 15-45 mg/day) leading up to enrollment.
* Karnofsky Performance Status ≥50%
* Adequate organ function, meeting all the following criteria within 30 days prior to enrollment:

  1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 × upper limit of normal (ULN)
  2. Total bilirubin ≤4 × ULN (≤8 × ULN in the setting of Gilbert's syndrome)
  3. Creatinine clearance (CrCl) ≥30 mL/min based on the Cockcroft-Gault formula
  4. Absolute neutrophil count ≥500/μL
  5. Prothrombin time (PT) or international normalized ratio (INR) ≤1.5 × ULN (unless prolonged due to therapeutic anticoagulation)
  6. Partial thromboplastic time (PTT) or activated PTT ≤1.5 × ULN (unless prolonged due to therapeutic anticoagulation)
  7. Platelet count ≥25 × 10^9/L (value must be obtained in the absence of platelet transfusion in the prior 7 days)
  8. Peripheral blasts <5%
* QT corrected by the Fridericia method (QTcF) ≤450 msec in males or ≤470 msec in females. Participants with QRS prolongation >100 msec may enroll if their QTcF is ≤480 msec. If QTcF is thought to be prolonged due to a modifiable factor (e.g., medication / electrolyte abnormality), QTcF may be reevaluated.
* Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test within 30 days prior to enrollment and a negative urine pregnancy test on Day 1 prior to randomization and dosing.
* WOCBP and male participants must agree to use a highly effective method of contraception starting at the first dose of trial therapy through 30 days after the last dose of trial therapy.

Key Exclusion Criteria

* Prior allogenic hematopoietic stem cell transplant (allo-HSCT) or solid organ transplant (other than corneal).
* Current use of systemic GCs for conditions other than VEXAS syndrome, which, in the opinion of the Investigator, would interfere with adherence to a GC taper regimen and/or assessment of efficacy.
* More than one prior admission to an intensive care unit due to a VEXAS Syndrome flare within the prior 6 months.
* Received ≥9 units of intensive red blood cell (RBC) transfusions in the 90 days prior to enrollment.
* Known concurrent myelodysplastic syndrome (MDS) requiring antineoplastic treatment, or allo-HSCT, or known high-risk or very high-risk MDS based on the Revised International Prognostic Scoring System (IPSS-R). Participants with MDS who do not meet these criteria may enroll.
* Malignancy within 1 year prior to enrollment with the exception of MDS (per exclusion criterion), curatively treated non-melanoma skin cancer, or curatively treated carcinoma in situ. Participants with pre-malignant hematologic conditions (e.g., monoclonal gammopathy of unknown significance [MGUS], clonal cytopenia of unknown significance) may enroll.
* Exposure to hypomethylating agents (HMA) within 6 months prior to enrollment, or exposure to more than 6 cycles of HMAs at any time.
* Exposure to non-GC anti-inflammatory therapy or hematologic support therapy within protocol defined timeframes prior to enrollment
* Exposure to anti-platelet therapy with the exception of low-dose aspirin (≤100 mg daily) within 28 days prior to enrollment.
* Known concomitant multiple myeloma, or serum M-protein ≥3 g/dL, involved-to uninvolved free light chain (FLC) ratio ≥100, or involved FLC level ≥100 mg/dL. Participants with MGUS may enroll.
* Systemic treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor or inducer within 5 half-lives prior to enrollment.
* Significant recent bleeding history defined as National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) grade ≥2 within 3 months prior to enrollment, unless precipitated by an inciting event.
* History of clinically significant cardiovascular disease, or clinically significant abnormalities in rhythm or conduction during Screening ECG, including:

  1. QT corrected by the Fridericia method (QTcF) > 480 msec within 30 days prior to enrollment; if QTcF is thought to be prolonged due to a modifiable factor (e.g., medication / electrolyte abnormality), QTcF may be re-evaluated
  2. Severe cardiac event (CTCAE grade ≥3) within 3 months prior to enrollment
  3. Heart failure resulting in limitations during ordinary activity.
* Arterial or venous thrombotic or embolic events, including deep vein thrombosis, pulmonary embolism, and cerebrovascular accident (including transient ischemic attacks), within 60 days prior to enrollment.
* Moderate or severe hepatic impairment that meets criteria for Child-Pugh Class B or C, or active viral hepatitis.
* Uncontrolled human immunodeficiency virus (HIV) off antiretrovirals, or on antiretrovirals with detectable viral load.
* Positive Quantiferon (or other interferon gamma release assay) during Screening.
* Known history of disseminated mycobacterial infection.
* Concurrent enrollment in another interventional trial, or treatment with an experimental therapy within 28 days or five half-lives prior to enrollment, whichever is longer.
* Pregnant, intending to become pregnant during the trial, or currently breastfeeding/lactating.
* Participants with any acute, active infection requiring systemic antimicrobial treatment at the time of enrollment. Exceptions are made for prophylactic antibiotics or chronic antibiotic therapy for non-acute conditions.
* Known hypersensitivity to pacritinib or any of the following inactive ingredients: microcrystalline cellulose, polyethylene glycol, and magnesium stearate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-05-22 (Estimated)

PRIMARY OUTCOMES:
Overall Clinical Response (OCR), defined as achieving Clinical Response or better at any time during the double-blind treatment period. | up to End of Week 24
  Difference in the proportion of participants achieving OCR for the pairwise comparison of pacritinib dose A vs. placebo and pacritinib dose B plus placebo vs. placebo

SECONDARY OUTCOMES:
Proportion of participants on each arm achieving each Best Response category (Clinical Biochemical Response, Clinical Response, Partial Clinical Response, Stable Disease, or Non-response). | up to End of Week 24
Number of flare-free days with GC dose <10 mg | up to End of Week 24
Hematologic Improvement - Erythroid | up to End of Week 24
  Erythroid (HI-E) at any time among participants with baseline hemoglobin <10 g/dL per modified International Working Group (IWG) criteria
Hematologic Improvement - Platelets | up to End of Week 24
  Platelets (HI-P) at any time among participants with baseline platelet count <100 × 10^9/L per modified IWG criteria
Change in health-related quality of life (QOL) as measured by Patient-Reported Outcomes Measurement Information Systems (PROMIS) fatigue short form | up to End of Week 24
  The PROMIS short form domains of fatigue 4a will be summarized, raw score from 4 to 20 (T-score from 33.7 to 75.8). A higher score is associated with more fatigue.
Change in health-related QOL as measured by PROMIS physical function short form | up to End of Week 24
  The PROMIS short form domains of physical function 4a will be summarized, raw score from 4 to 20 (T-score from 22.5 to 57.0). A higher score is associated with better physical function.
Change in health-related QOL as measured by PROMIS sleep disturbance short form | up to End of Week 24
  The PROMIS short form domains of sleep disturbance 4a will be summarized, raw score from 4 to 20 (T-score from 32.0 to 73.3). A higher score is associated with more sleep disturbance.
Change in health-related QOL as measured by the 36-item short form (SF) Survey | up to End of Week 24
  The SF-36 Survey measures eight domains of health status; physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health. The values for each domain range from 0 to 100, with the higher score indicating a better health status.
Change in health-related QOL as measured by Patient's Global Impression of Change (PGIC) response | up to End of Week 24
  The number and percentage of participants achieving PGIC response (reporting symptoms as "much" or "very much" improved).
Mean plasma concentration of pacritinib | up to Week 24 (pre-dose only)
  Mean plasma concentrations (pre-dose and post-dose) will be determined for each pharmacokinetic sampling timepoint.
Change in pharmacodynamic (PD) inflammatory biomarker: C-reactive protein (CRP) | up to 30-day Post-End of Trial
Change in PD inflammatory biomarker: erythrocyte sedimentation rate (ESR) | up to 30-day Post-End of Trial
Change in PD inflammatory biomarker: ferritin | up to 30-day Post-End of Trial

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — Sobi, Inc.
Locations (40):
- United States (10):
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - University of Maryland Medical Center Midtown Campus, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - Cleveland Clinic - Cleveland, Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - UT MD Anderson Cancer Center, Houston, Texas
  - University of Utah Healthcare, Salt Lake City, Utah
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Canada (4):
  - Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hospital du Sacre-Coeur in Montreal, Montreal, Quebec
- France (6):
  - Lille University Hospital Center, Lille
  - Saint-Antoine Hospital - APHP, Paris
  - Tenon Hospital - APHP, Paris
  - Hospices Civils de Lyon - Lyon Sud, Pierre-Bénite
  - University Hospital Center of Poitiers, Poitiers
  - IUCT-Oncopole, Toulouse
- Germany (6):
  - University Hospital Tuebingen, Medical Clinic II, Hematology, Oncology, Clinical Immunology and Rheumatology, Tübingen, Baden-Wurttemberg
  - Hospital Rechts der Isar of the Technical University of Munich, Clinic and Polyclinic for Internal Medicine III: Hematology and Internal Oncology, Munich, Bavaria
  - University Hospital Hamburg-Eppendorf, Hamburg, Hamburg
  - University Hospital Duesseldorf, Düsseldorf, North Rhine-Westphalia
  - University Hospital Carl Gustav Carus Dresden, Medical Clinic and Polyclinic I, Dresden, Saxony
  - University Hospital Schleswig-Holstein, Lübeck, Schleswig-Holstein
- Italy (4):
  - Hospital San Raffaele, IRCCS, Unit of Immunology, Rheumatology, Allergy and Rare Diseases, Milan
  - University Hospital of Padova, Rheumatology Unit, Department of Medicine - DIMED, Padua
  - AUSL of Reggio Emilia - Hospital Arcispedale S. Maria Nuova, Complex Structure of Rheumatology, Reggio Emilia
  - Foundation PTV - Polyclinic Tor Vergata Biomedicine and prevention, Roma
- Japan (3):
  - Fukushima Medical University Hospital, Fukushima
  - Nagasaki University Hospital, Nagasaki
  - Yokohama City University Hospital, Yokohama
- Spain (3):
  - Hospital Clinic of Barcelona, Barcelona
  - Catalan Institute of Oncology, Hospital Duran i Reynals, Department of Clinical Hematology, L'Hospitalet de Llobregat
  - University Clinical Hospital of Salamanca, Salamanca
- United Kingdom (4):
  - St James's University Hospital, Leeds
  - Royal Free Hospital, London
  - King's College Hospital, Department of Hematology, London
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related trial documents. Patient level data will be anonymized and trial documents, if applicable will be redacted to protect the privacy of trial participants.
URL: https://www.sobi.com/en/policies